CLINICAL TRIAL: NCT06966505
Title: Patients Admitted to ICU After a Suicide Attempt: Physical and Mental Symptoms and the Patients' Experiences With Treatment
Brief Title: Patients Admitted to ICU After a Suicide Attempt
Acronym: SA_ICU
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Kristin Hofsø, Professor, Oslo University Hospital
Other Study IDs: 202196; REK (Other: Regional Etisk Komite)
Record Dates: First submitted 2025-04-11; First posted 2025-05-12 (Actual); Last update posted 2025-05-12 (Actual); Status verified 2025-05

CONDITIONS: Suicide Attempt
Keywords: Suicide attempters in ICU; ICU
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients that has been admitted to the ICU after a suicide attempt: We have only included suicide attempters that have been admitted to an ICU

SUMMARY:
The goal of this study is to increase the knowledge on the experience and symptom profile to suicide attempters admitted to an ICU.

Suicide is one of the most frequent causes of death in young age groups in Norway, and the rates has not decreased in Norway in 20 years despite governmental and health care actions when it comes to prevention, knowledge and treatment. The medically most serious suicide attempts need treatment in intensive care units (ICU). In addition, being an ICU patient is associated with the experience of several traumatic events and symptoms related to treatment. These experiences often have a negative impact on their quality-of-life post discharge. In addition, patients who have tried to end their life often have experienced negative life events prior to the suicide attempt.

A systematic review conducted on attitudes towards people who self-harm, pointed out inappropriate staff behaviour, lack of patient-involvement, poor knowledge among the health care professionals and issues with aftercare to this particular patient group. Healthcare personnel are important stakeholders in suicide prevention, but they can experience lack of confidence when caring for suicidal patients and negative attitudes have an impact on access to treatment. Building knowledge addressing mental health stigma and negative attitudes is possible with training and education.

As there are little evidence regarding the experience, symptom profile and the follow up for this specific sub-group of the ICU population, this project aims to investigate three aspects affecting the suicide attempt patient in the ICU; First, the symptom burden of suicide attempt patients experienced both in the ICU and post-discharge during 6 months will be examined. Second, the ICU nurses' attitudes towards the suicide attempt patient will be explored. Finally, after ICU discharge the patients feeling of hopelessness and other symptoms will be investigated, and the general experience as an ICU patient. This project is highly innovative and will fill a significant gap in knowledge.

DETAILED DESCRIPTION:
In this project patients will be included as soon as possible after the ICU admission. A research nurse trained for t inclusion of this specific patient population will ask the patient for inclusion, after a physician or psychiatrist have defined the cause of admission as a suicide attempt. Patients will be asked to fill out questionnaires in the ICU, facilitated by the study nurse if they consent to study participation, and then again after 3 and 6 months.

Patients with medically serious suicide attempts have a higher risk of suicide than others. We know that half of the population of patients dying of suicide have previously self-harmed, and that the rate of suicide in the self-harm population is approximately 100 times higher than the general population.

It is often unclear whether the reason behind the suicide attempt was an explicit wish to die or an act of deliberate self-harm (DSH) where the patient was coping with psychological pain but had no wish to die. The vast majority of previous research on suicidal patients has used the definition of deliberate self-harm when including patients. These two groups of patients are described as overlapping, where risk factors for later suicide are common, and self-destructive behavior is important. In an acute setting, when medical treatment is in focus, the intention is rarely evaluated, mainly because the poisoning or treatment of hanging and shooting reduces consciousness. All patients treated for suicide attempt in the ICU will therefore be included, and their suicidal intent will be evaluated after inclusion.

Previous research has described 5 key symptoms that should be evaluated every day in ICU patients, and includes pain, thirst, anxiety, dyspnea and tiredness. Only one older study has been identified to address symptoms and experiences by suicide attempt patients in the ICU, and patients from this study described experiences of pain, despair, shame and guilt.

The attitudes towards suicide of the ICU personnel may affect the care provided, and also the life after discharge for the patient. Hopelessness is one of the strongest predictors for suicide and repeated self-harm. Hopelessness is recommended and commonly used as assessment in the context of suicidal behaviour. Besides its crucial role in suicidality, hopelessness is an important construct in the context of life satisfaction, compliance and recovery in medical care.

The general suicide attempt patient-group have increased short -and long-term mortality of both suicide and natural deaths compared to the general population and thus underlines the importance of structured follow-up. The negative consequences of surviving an ICU stay have received increased attention in recent years, as decreased mortality rates have contributed to a high number of ICU Survivors. The identification of post-intensive care Syndrome (PICS) has been of great importance for increasing awareness about health issues in ICU survivors. PICS conceptualizes health challenges within physical, psychological and cognitive domains of health. However, PICS needs to be addressed and investigated in the suicide attempt population admitted to ICU as well, as descriptions of this specific population does not seem to exist.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have attempted suicide, and
* patients ≥18 years, and
* have been ≥12hours in the ICU
* suicide attempt have been defined as "a potentially self-injurious behaviour with a non-fatal outcome, for which there is evidence (either explicit or implicit) that the person intended at some (non-zero) level to end their lives. A suicide attempt may or may not result in injuries". All suicide methods leading to hospitalization are included (hanging, drowning, jump/ fall from heights, shooting, self-poisoning, cutting and other methods), as defined in International classification of diseases version 10 (ICD-10, chapter X)
* trained research personnel from the research group will conduct the evaluation with the medical team treating the patient to identify the suicide attempt patient

Exclusion Criteria:

* Not able to read or understand Norwegian
* Patients with no permanent address in Norway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to an ICU after a suicide attempt.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Symptoms | Day 1 in the ICU (or first possible day to self-report), and at 3 and 6 months after ICU admission.
  Symptoms will be measured using Patients Symptom Survey (10 symptoms), and is a multi-dimensional symptom Assessment Scale developed for the ICU population.

SECONDARY OUTCOMES:
Hopelessness | Day 1 in the ICU (or first possible day to self-report) and at 3 and 6 months after ICU admission
  Will be measuerd using Bechs hopelessness scale. It has a range from 0 (no hopelessness) to 20 (maximum hopelessness).

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Departement, Oslo, Oslo County, Norway